CLINICAL TRIAL: NCT00480350
Title: RiSolubles™, the Soluble Fraction of Rice Bran for HIV-Infected Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: shah1HMO-CTIL
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-03

CONDITIONS: HIV Infections
Keywords: HIV; virological response; CD4; food supplement; Human Immunodeficiency Virus; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: rice based food supplement

SUMMARY:
HIV infection is a growing problem in Israel with over 4000 known patients who are either infected with the virus or have developed AIDS. Patients are usually followed for years until they develop an increase in their viral load (HIV-1 RNA) or their CD4 + cells decline. At this point, patients are usually treated with Highly Active, Anti-Retroviral Therapy (HAART). The mainstay of response to such treatment is the lowering of viral load and increase in CD4+ cells. Food supplements for HIV patients have been given in several studies, with controversial results. A meta-analysis published recently [1] assessed whether micronutrient supplements are effective in reducing morbidity and mortality in adults and children with HIV infection. They recommended supporting the current WHO recommendations to promote and support adequate dietary intake of micronutrients wherever possible. We expect to enroll 140 subjects in this randomized, double blind, placebo controlled study. Seventy subjects will be enrolled in the rice-supplement arm and 70 subjects in the control group, which will receive supplemental, flavored dextrose to their current medical treatment. The treatment duration is 24 weeks with follow-up at 36 weeks from enrollment. The target population is HIV-1 infected individuals who may be either on anti-retroviral therapy or not on therapy. Subjects must be with either CD4+ cells are <500 cells/mm3, or HIV plasma RNA level is > 5000 copies/ml. The primary objective is to demonstrate the efficacy of food supplementation versus a flavored-dextrose supplement with respect to increment of patient CD4+ cell count from baseline at 24 weeks, or virological response defined as lowering of plasma HIV-1 RNA and immunologic response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented HIV-1 infection
* Male and female ages > 18 years old
* Subjects who have given informed consent
* Subjects may either receive or not receive antiretroviral therapy at the time of enrollment
* Plasma HIV-1 RNA higher than 5000 copies/ml
* OR
* Patient CD4+ cell count less than 500 cells/mm3
* Patients who can comply with protocol requirements

Exclusion Criteria:

* Patients incapable of oral intake
* Patients who are allergic to rice
* Pregnant or breast-feeding women
* Active drug abuse which, in the opinion of the investigator, is expected to interfere with the subject's ability to adhere to the study procedures
* Active, clinically-significant disease or life-threatening disease that would compromise the subject's safety or outcome of the study
* Any medical or psychiatric condition which, in the opinion of the investigator, could compromise the subject's safety or adherence to the trial protocol
* Patients who have started their anti-HIV treatment within less than 3 months from inclusion in the study. However, patients who have changed anti-HIV medication but have initiated therapy more than 3 months before inclusion will be eligible for the study.
* Patients known to suffer from diabetes mellitus
* Participation in any other clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-09; Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be an increment of CD4+ cells by a mean of 25% or increase of 100 cells/ mm3 at week 24 in the treatment group | 24 weeks

SECONDARY OUTCOMES:
The proportion with virologic response defined as a plasma HIV-1 reduction of 1 log at week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allon E Moses, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel